CLINICAL TRIAL: NCT00585143
Title: Pharmacokinetics of ABT-335 and Rosuvastatin in Subjects With Normal Renal Function and Renal Impairment
Brief Title: Safety Study to Evaluate the Effects of Mild and Moderate Renal Impairment on the Pharmacokinetics of ABT-335 and Rosuvastatin When Administered Concomitantly
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M10-070
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Dyslipidemia, Renal Insufficiency
Keywords: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias; Renal Insufficiency | interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-335; Drug: Rosuvastatin

INTERVENTIONS:
Drug: ABT-335 — 45 mg once daily for 10 consecutive days
Drug: Rosuvastatin — 10 mg once daily for 10 days

SUMMARY:
Safety Study to Evaluate the Effects of Mild and Moderate Renal Impairment on the Pharmacokinetics of ABT-335 and Rosuvastatin When Administered Concomitantly

ELIGIBILITY:
Inclusion Criteria

Body Mass Index (BMI) 19 to 33, inclusive

Either normal kidney function, or mild or moderate kidney impairment

Exclusion Criteria

Use of any medications, vitamins and/or herbal supplements within 2 weeks prior to study drug administration, except those required for management of renal disease.

History of epilepsy, any clinically significant cardiac, respiratory, renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of the active ingredients and metabolites of ABT-335 and rosuvastatin | Days 1, 8, 9, and 10

SECONDARY OUTCOMES:
Safety and tolerability of the study drugs | Study duration

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (6):
- United States (6):
  - Site Reference ID/Investigator# 6610, Gainesville, Florida
  - Site Reference ID/Investigator# 6738, Miami, Florida
  - Site Reference ID/Investigator# 7723, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 7319, Knoxville, Tennessee
  - Site Reference ID/Investigator# 6928, San Antonio, Texas
  - Site Reference ID/Investigator# 8280, Richmond, Virginia